CLINICAL TRIAL: NCT01823939
Title: Two-Part, Single-Centre Pharmacokinetic Study of iOWH032 in Adult Male and Female Healthy Volunteers, and Adult Males With Cholera
Brief Title: PK Study of iOWH032 in Adult Male/Female Healthy Volunteers & Adult Males With Cholera
Acronym: PISCES
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PK Study; DDP CFT PO 201 (Other Grant/Funding Number: Bill & Melinda Gates Foundation)
Record Dates: First submitted 2013-03-27; First posted 2013-04-04 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Diarrhea; Cholera
Keywords: Cholera; V. Cholerae O1; iOWH032; diarrhoea; pharmacokinetic; Bangladesh
MeSH Terms: conditions — Diarrhea; Cholera | interventions — IOWH-032

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Males / Females (Healthy) (Other): Part A: This initial part of the study will be conducted in adult Bangladeshi healthy volunteers (4 males, 4 females) to assess the pharmacokinetics, safety, and tolerability of single doses of iOWH032. Participants will be admitted to the Clinical Trial Unit (CTU) of icddr,b (located at a 10 minute drive from the icddr,b main campus) the day prior to dosing and remain for 48 hours after dosing, unless treatment and/or follow-up of an adverse event (AE) require longer in-unit observation or treatment.
  Interventions: Drug: iOWH032
- Males (Patient) (Other): Part B: Patients will be eligible for the study if they have clinically severe dehydration and meet all other inclusion and exclusion criteria. Upon signing consent, they will be admitted to the Research Ward of the Dhaka Hospital of icddr,b.
  Interventions: Drug: iOWH032

INTERVENTIONS:
Drug: iOWH032 — Part A: Participants will be randomized at a 3:1 ratio to receive treatment with iOWH032 or placebo. A randomisation code will be generated. Each participant will be assigned the next participant number available and thereby will be assigned randomly. Active treatment will consist of an oral tablet containing 300 mg of iOWH032. The placebo will consist of identical looking tablets.
  Part B: There will be no randomization during this trial. All eligible patients will receive 300 mg of iOWH032.

SUMMARY:
This study will assess if the pharmacokinetics, safety and tolerability of iOWH032 are grossly different in 1) Bangladeshi healthy population and 2) Bangladeshi cholera patients. This is not a hypothesis-driven research study.

DETAILED DESCRIPTION:
This study will be conducted in two parts.

The first part (Part A) will evaluate the pharmacokinetics, safety and tolerability of iOWH032 in healthy, adult Bangladeshi volunteers.

The second part (Part B) will evaluate the pharmacokinetics, safety and tolerability of iOWH032 in adult Bangladeshi patients with cholera. While female participants will be included in Part A, only male patients will be enrolled in Part B. The rationale for excluding women in Part B is the difficulty in separating urine from stool in severely dehydrated females with rapid rates of purging. Moreover, it has been difficult to retain adult females in the hospital after improvement of their diarrhoea because of their household responsibilities, which might impact compliance in this small study. Further, no sex differences in the pharmacokinetics of iOWH032 were found in the study conducted in healthy subjects in the US, which included 42 males and females, nor have sex differnces been observed in preclinical studies.

ELIGIBILITY:
INCLUSION CRITERIA - Part A:

An individual will be considered eligible for participation in the trial if the following inclusion criteria are satisfied:

1. Male or female between 18 and 55 years, inclusive;
2. Female participants are non-pregnant and non-lactating. Female participants of childbearing potential (including perimenopausal women who had menstrual bleeding within the past two years) must use appropriate birth control (abstinence and/or double barrier methods) for 30 days after dosing. Acceptable double barrier methods are the following forms of contraception: condom, contraceptive sponge, hormonal contraceptives, intrauterine devices, and diaphragm or cervical ring with spermicidal gel or foam. Women are considered to be not of childbearing potential if they have been surgically sterilized (physician-documented hysterectomy, bilateral oophorectomy or bilateral tubal ligation). All female participants must have a negative pregnancy test at screening and on admission to the CTU.
3. Written informed consent for participation in the study.

INCLUSION CRITERIA - Part B:

A patient will be considered eligible for participation in the trial if the following inclusion criteria are satisfied on admission (Day 1) to the hospital:

1. Males aged 18 years to 55 years, inclusive;
2. Duration of illness: History of acute watery diarrhoea of less than 24 hours duration without fever or visible blood in faeces;
3. Clinical signs and symptoms of severe dehydration;
4. A stool Dark-field microscopy or Rapid Strip test demonstrating presence of V. cholerae.
5. Written informed consent for participation in the study.

EXCLUSION CRITERIA - Part A:

An individual with any of the following criteria at screening for study enrolment will not qualify for the study:

1. Evidence or history of clinically significant allergic, haematological, immunological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease; or any other condition likely to interfere with the absorption, disposition, metabolism, or excretion of the investigational product;
2. History of cancer with the exception of basal cell or squamous cell (skin) carcinoma;
3. History of drug or alcohol abuse or dependence (based on DSM-IV criteria) within the past two years;
4. Donated blood or plasma, or experienced significant loss of blood within eight weeks prior to admission to the CTU or who plan to donate blood or plasma within one month after study participation;
5. Sustained systolic blood pressure > 140 mmHg or < 95 mmHg or a diastolic blood pressure > 95 mmHg obtained in the seated position;
6. Heart rate at rest of < 40 bpm or > 100 bpm;
7. Clinically significant abnormal ECG findings, as determined by the investigator;
8. Clinically significant abnormal laboratory test results, as determined by the investigator;
9. Currently uses or has used tobacco or nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, etc.) within 30 days prior to admission to the CTU;
10. Evidence or history of any clinically significant illness as per the Investigator's discretion
11. Past history of gastric, small intestinal, or colonic surgery, not including appendectomy or cholecystectomy;
12. Positive HBsAg or anti-HCV Ab;
13. Positive urine test for drug(s) of abuse: benzodiazepines, cocaine, marijuana, methamphetamine, and opiates;
14. Known hypersensitivity to, or intolerance of the excipients in the study medication;
15. Taken over-the-counter (OTC) or prescription medications or herbal supplements (other than hormonal contraceptives, acetaminophen and/or multivitamins [acetaminophen 2gm/day and multivitamins allowed up to 48 hours prior to dosing]) within 14 days;
16. Participants unwilling or unable to take part in this study or refusing to sign informed consent;
17. Participants previously enrolled in this or any other investigational study with the past 30 days.
18. Any current or past condition or laboratory abnormality, which, in the opinion of the investigator, could confound or interfere with evaluation of safety, tolerability, and/or pharmacokinetics of the investigational drug, or prevent compliance with the study protocol.

EXCLUSION CRITERIA - Part B:

A patient with any of the following criteria at screening for study enrolment will not qualify for the study:

1. History of receiving antimicrobial or anti-diarrhoeal medication (loperamide, diphenoxylate, etc.) within the seven days of admission;
2. Clinically significant abnormal ECG findings, with the exception of sinus tachycardia, premature atrial contractions, or ECG intervals within normal limits for sinus rate;
3. Use of drugs metabolized predominantly via CYP2C93 within seven days of admission;
4. Evidence or history of any clinically significant illness as per the Investigator's discretion
5. Evidence or history of concomitant infection requiring antimicrobial therapy
6. Known hypersensitivity to, or intolerance of iOWH032 or the excipients
7. Past history of gastric, small intestinal, or colonic surgery, not including appendectomy or cholecystectomy
8. Patients unwilling or unable to take part in this study or refusing to sign informed consent
9. Patients previously enrolled in this or any other investigational study with the past 30 days.
10. Any current or past condition or laboratory abnormality, which, in the opinion of the investigator, could confound or interfere with evaluation of safety, tolerability, and/or pharmacokinetics of the investigational drug, or prevent compliance with the study protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Calculation of concentration-time data | Day 1 through end of treatment (Day 150)
  For both Part A and Part B:
  * pharmacokinetic parameters
  * adverse events (AEs)
  * laboratory values
  * physical examination and vital sign findings
  * summary statistics
  For Part B, patients with culture-proven V. cholerae O1 infection will be evaluated independently of those with a negative culture. Those who are culture negative for V. cholerae but have received iOWH032 will remain in the study and the same protocol will be followed for their management including the follow up visit.

SECONDARY OUTCOMES:
Measure of Adverse Events | 7 days after receipt of the single dose
  The safety and tolerability endpoint for this study is adverse events (AEs). All participants and patients receiving investigational product (iOWH032) will be included in the safety analysis. Laboratory values, physical examinations and vital signs will be summarized over time and treatment group using the descriptive statistics and plots.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Salam, MBBS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Dhaka Hospital - icddr,b (International Centre for Diarrhoeal Disease Research, Bangladesh), Mohakhali, Dhaka Division, Bangladesh